CLINICAL TRIAL: NCT07291531
Title: Optimizing Pulp Management Strategies for Autotransplantation of Fully Developed Third Molars: A Three-Arm Randomized Controlled Trial
Brief Title: Optimizing Pulp Management in Autotransplantation of Mature Third Molars: A Randomized Controlled Trial
Acronym: OPuM-ATM3
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-1392
Record Dates: First submitted 2025-12-07; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Tooth Avulsion; Dental Pulp Diseases; Tooth, Impacted
Keywords: Autotransplantation; Third molar; Root canal therapy; Apical surgery; Root-end resection; mature tooth
MeSH Terms: conditions — Tooth Avulsion; Dental Pulp Diseases; Tooth, Impacted

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Postoperative Root Canal Therapy (PRCT) (Active Comparator): Participants in this group will receive conventional autotransplantation of a fully developed third molar. No additional apical procedure is performed on the donor tooth during surgery. Standard non-surgical root canal therapy will be initiated and completed within 2-4 weeks after the transplantation procedure.
  Interventions: Procedure: Postoperative Root Canal Therapy
- Apical Surgery with Retrograde Filling (AS) (Experimental): Participants in this group will receive autotransplantation of a fully developed third molar with intraoperative apical surgery. During surgery (ex vivo), the root apex (approximately 3mm) of the donor tooth is resected, followed by retrograde cavity preparation and obturation with a biocompatible material (e.g., MTA). Standard non-surgical root canal therapy will also be initiated and completed within 2-4 weeks postoperatively.
  Interventions: Procedure: Intraoperative Apical Surgery with Retrograde Filling
- Root-End Resection Only (RER) (Experimental): Participants in this group will receive autotransplantation of a fully developed third molar with intraoperative root-end resection only. During surgery (ex vivo), the root apex (approximately 3mm) is resected to enlarge the apical foramen, but no retrograde preparation or filling is performed. No prophylactic root canal therapy is planned postoperatively. Remedial root canal therapy will be provided only if signs/symptoms of pulp necrosis or apical periodontitis develop during follow-up.
  Interventions: Procedure: Intraoperative Root-End Resection

INTERVENTIONS:
Procedure: Postoperative Root Canal Therapy — This intervention involves the standard non-surgical root canal treatment of the autotransplanted tooth. It is performed after the surgical transplantation procedure, typically initiated within 2-4 weeks postoperatively. The procedure includes pulp extirpation, biomechanical preparation, disinfection, and obturation of the root canal system using standard techniques and materials (e.g., gutta-percha and sealer).
  Other Names: PRCT
  Arms: Postoperative Root Canal Therapy (PRCT)
Procedure: Intraoperative Apical Surgery with Retrograde Filling — This surgical intervention is performed on the donor tooth during the transplantation procedure, while the tooth is outside the mouth (ex vivo). It consists of: 1) Resection of approximately 3mm of the root apex; 2) Preparation of a retrograde cavity at the resected apex; and 3) Obturation of this cavity with a biocompatible material, such as Mineral Trioxide Aggregate (MTA), to achieve a seal. This is followed by postoperative root canal therapy (as described in Intervention 1).
  Other Names: AS
  Arms: Apical Surgery with Retrograde Filling (AS)
Procedure: Intraoperative Root-End Resection — This surgical intervention is performed on the donor tooth during the transplantation procedure, while the tooth is outside the mouth (ex vivo). It involves the resection of approximately 3mm of the root apex only, with the aim of enlarging the apical foramen. Crucially, no retrograde preparation or filling is performed. Postoperatively, no prophylactic (preventive) root canal therapy is planned. The goal is to promote revascularization and survival of the pulp. Remedial root canal therapy is provided only if clinical or radiographic signs of pulp necrosis or apical periodontitis develop during follow-up.
  Arms: Root-End Resection Only (RER)

SUMMARY:
This study aims to find the best way to use your own healthy wisdom tooth to replace the bad tooth. After transplantation, how to manage the "tooth nerve" (dental pulp) inside the tooth is a key question. Currently, doctors have three different management strategies, but it is not clear which one is most beneficial for long-term success.

This study will compare these three strategies:

Performing standard root canal treatment (removing the tooth nerve) a few weeks after transplantation.

Performing a special procedure to treat and fill the root tip during the transplant surgery, followed by root canal treatment later.

Simply trimming the root tip during the transplant surgery, hoping to preserve the vitality of the tooth nerve and thereby avoid subsequent root canal treatment.

If you agree to participate, you will be randomly assigned to one of these groups to receive treatment. Afterwards, we will need to schedule regular check-ups for you over a period of 5 years (including X-rays and examinations) to monitor the healing of the transplanted tooth, check for any problems, and assess the status of the tooth nerve.

Your participation will help us identify the most effective and long-lasting treatment method, thereby benefiting future patients in similar situations.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-40 years.
2. Requires extraction of a non-restorable first or second molar AND possesses a fully developed, morphologically healthy ipsilateral third molar as a donor tooth.
3. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Presence of acute infection or insufficient bone volume at the recipient site.
2. Donor tooth exhibits caries, periapical pathology, or periodontal disease.
3. Uncontrolled systemic disease (e.g., diabetes, immunosuppression), pregnancy, or lactation.

   Smoking habit of >10 cigarettes per day.
4. Inability or unwillingness to comply with the long-term follow-up schedule.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 360 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2031-06 (Estimated); Study Completion 2032-06 (Estimated)

PRIMARY OUTCOMES:
Success Rate | 1 year and 5 years postoperatively
  Comprehensive success defined as the transplanted tooth being present, functional, asymptomatic (no pain on percussion, no sinus tract), with healthy gingiva, and no radiographic evidence of progressive inflammatory root resorption or periapical radiolucency.
Survival Rate | 1 year and 5 years postoperatively
  The proportion of transplanted teeth remaining in the oral cavity and functional.
Incidence of Inflammatory Root Resorption | 1 year and 5 years postoperatively
  The proportion of transplanted teeth exhibiting radiographic signs of inflammatory root resorption (periapical radiolucency adjacent to the root surface with loss of lamina dura) on periapical radiograph or CBCT.

SECONDARY OUTCOMES:
Pulp Revascularization/Survival (RER Group) | Postoperative 3, 6, 12 months, and then annually up to 5 years
  Assessment of pulp vitality via clinical tests (electric pulp test, cold test) in the RER group.
Radiographic Periodontal Ligament Healing | Postoperative 3, 6, 12 months, and then annually up to 5 years
  Evaluation of the uniformity, continuity, and width of the periodontal ligament space on periapical radiographs/CBCT at specified intervals, and detection of ankylosis.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD will be shared with researchers upon reasonable request and approval of a proposal.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The IPD and supporting documents will become available 12 months after the publication of the primary results** (the manuscript reporting the primary outcomes). They will remain accessible for at least 5 years.
Access Criteria: Access will be granted to researchers who provide a methodologically sound proposal, approved by an independent review committee ("data access committee"). Proposals should be directed to the corresponding author. Requestors will need to sign a data access agreement specifying that data will be used only for the approved purpose, not to attempt to identify participants, and will be destroyed after use.